CLINICAL TRIAL: NCT06331754
Title: Technology-Enabled Remote Hypertension Management To Advance Health Equity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atman Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATMANHEALTH001
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: non-blinded pragmatic cluster-randomized controlled trial with a single intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-enabled blood pressure management (Experimental): The intervention will consist of a technology-enabled remote hypertension management program. Participants will be given a cellular blood pressure (BP) cuff and patients with heart failure and chronic kidney disease stage 3b-5 will be given a scale also. Patients will undergo a series of protocolized software-driven medication initiation and titration steps until they reach a blood pressure target of systolic blood pressure < 130 mmHg and diastolic blood pressure < 80 mmHg. Patients will be subsequently monitored for up to 12 more months. If their blood pressure increases, they can re-enter active management.
  Interventions: Other: Technology-enabled blood pressure management
- No intervention (No Intervention): Patients meeting inclusion care undergoing usual care in control clinics.

INTERVENTIONS:
Other: Technology-enabled blood pressure management — The intervention will consist of a technology-enabled remote hypertension management program.
  Arms: Technology-enabled blood pressure management

SUMMARY:
The primary objective of this study is to reliably estimate the difference in blood pressure control of a technology-enabled solution for blood pressure (BP) management over usual care. The study will also assess patient and provider satisfaction with the solution. Finally, the investigators will estimate the economic impact of the intervention in terms of resource utilization.

DETAILED DESCRIPTION:
The study design is a non-blinded pragmatic cluster-randomized controlled trial with a single intervention. Participants with uncontrolled hypertension will be identified from a randomly selected group of primary care clinics. Participants from half of the clinics will be enrolled in the intervention arm while the others will receive usual care. Participants in the intervention arm will undergo a series of software-driven medication initiation and titration steps until they reach a blood pressure target of systolic blood pressure < 130 mmHg and diastolic blood pressure < 80 mmHg. Participants will be subsequently monitored for up to 12 more months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years - 100 years
* uncontrolled hypertension: as defined as SBP > 140 or DBP > 90 on 2 successive clinic visits

Exclusion Criteria:

* hearing impaired
* visually impaired
* cognitively impaired
* hospice care
* on hemodialysis at enrollment
* New York Heart Association Class IV heart failure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-18 (Estimated); Primary Completion 2025-09-17 (Estimated); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Difference in SBP change | 6 months after enrollment
  Difference in mean change in systolic blood pressure (SBP)

SECONDARY OUTCOMES:
HEDIS proportion | 6 months after enrollment
  Difference in the proportion of patients meeting HEDIS definition of controlled hypertension (SBP < 140 AND DBP < 90) between intervention and usual care: overall and by patient group and by age, race, sex strata
Difference in DBP change | 6 months after enrollment
  Difference in mean change in diastolic blood pressure (DBP)

OTHER OUTCOMES:
Home measured change in SBP and DBP | 6 months
  Home measured change in blood pressure in intervention group - more accurately measured: overall and by patient group
Patient satisfaction | 6 months
  A patient satisfaction survey with questions similar to the Consumer Assessment of Healthcare Providers and Systems will be used.
Provider satisfaction | 6 months
  A survey instrument will be developed and administered to assess provider satisfaction with having a remote team manage their patients.
Mean time required per patient for provider | 6 months
  Cumulative time in minutes for all interactions, including documentation.
Mean time required per patient for navigator | 6 months
  Cumulative time in minutes for all interactions, including documentation.
Proportion of patients measuring blood pressure at directed frequency | 6 months
  Proportion of patients measuring blood pressure at least twice a day during active management period.
Resource utilization | 18 months
  Difference in resource utilization between intervention and usual care for different patient groups using claims data.

IPD SHARING:
Plan to Share IPD: Undecided